CLINICAL TRIAL: NCT01230619
Title: A Two Day, Randomised, Single Blind, Parallel Group Trial of Repeat Doses of Intranasal RV568 in the Vienna Challenge Chamber in Subjects With Seasonal Allergic Rhinitis (SAR)
Brief Title: Vienna Challenge Chamber Study Using RV658 in Subjects With Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Respivert Ltd (Industry)
Responsible Party: Dr Garth Rapeport, Respivert Ltd
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RVH002; 2010-022113-25 (EudraCT Number)
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- RV568 treatment group (Experimental)
  Interventions: Drug: RV568
- Placebo treatment group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RV568 — RV568 400 ug administered as nasal drops twice daily on Day 1, RV568 800 ug administered as nasal drops once daily on Day 2
  Arms: RV568 treatment group
Drug: Placebo — Placebo administered as nasal drops twice daily on Day 1, Placebo administered as nasal drops once daily on Day 2
  Arms: Placebo treatment group

SUMMARY:
RV568 is being developed for the treatment of diseases such as asthma, COPD and allergic rhinitis (e.g. hayfever). The main aim of this study is to investigate whether RV568 ameliorates the nasal symptoms to low doses of grass pollen in healthy subjects with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy
* History of seasonal allergic rhinitis
* Male aged between 18 and 55 years
* Body weight >/= 50 kg with BMI in range 19 - 29 kg/m2 (inclusive)
* Exhibits a moderate response to 4 hour exposure to grass pollen in the challenge chamber with a total nasal symptom score (TNSS) of >/= 6
* Positive skin prick test (wheal >/= 4 mm) for grass pollen
* Positive total IgE result (RAST class >/= 2) for grass pollen
* Current non-smoker who has not used tobacco in the past 6 months with a pack history of </= 10 pack years
* Baseline FEV1 >/= 80% and FEV1/FVC >/= 70% of predicted values
* No conditions or factors that may preclude subjects ability to remain in the challenge chamber for a period of 6 hours
* capable of giving informed consent and is compliant with protocol requirements
* available to complete all study measurements

Exclusion Criteria:

* structural nasal abnormalities or nasal polyps, history of frequent nosebleeds, recent nasal surgery or recent (within 3 weeks) or ongoing upper respiratory tract infection
* history of drug allergy
* participation in another clinical trial or has participated in a study using an NCE within the previous 3 months, or any clinical study within 1 month
* taking regular (or a course of) medication whether prescribed or not, including steroids, vitamins, macrolides, anti-fungal agents and herbal remedies. Paracetamol (</= 2g / day) and occasional short acting beta agonists are permitted
* use of oral, injectable or dermal steroids within 5 weeks or intranasal and/or inhaled steroids within 1 week of the screening visit
* past or present disease, which as judged by the investigator, may affect the outcome of the study
* regular consumption of > 21 units alcohol per week
* infected with Hepatitis B, Hepatitis C, or HIV virus
* current or chronic history of liver disease, or known hepatic or biliary abnormalities
* positive test for drugs of abuse or alcohol at screening
* previously known allergy to any of the active or inactive ingredients in the study medication
* mentally or legally incapacitated
* any other reason that the investigator considers makes the subject unsuitable to participate

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Total nasal symptom score (TNSS) | 2 day treatment period
  Nasal congestion, rhinorrhoea, nasal itching and sneezing will be scored on a categorical scale from 0 to 3. Individual scores will be summed to produce the TNSS

SECONDARY OUTCOMES:
Eye symptom score | 2 day treatment period
  Watery eyes, itchy eyes, red eyes will be scored on a categorical scale of 0 to 3
Global symptom score | 2 day treatment period
  Sum of symptom scores; TNSS, Eye symptom score, Other symptom score,(comprising congestion, rhinorrhoea, nasal itching, sneezing, watery eyes, itchy eyes, red eyes, cough, itchy throat and itchy ears) will be scored categorically from 0 to 3
Nasal airflow resistance | 2 day treatment period
Safety parameters | 3 weeks
  Spirometry, 12-lead ECG, laboratory assessments and adverse event assessment

CONTACTS AND LOCATIONS:
Overall Officials: Prof Dr Friedrich Horak, MD, Principal Investigator — Institute for Allergy Research - Vienna Challenge Chamber
Locations (1):
- Institute for Allergy Research, Vienna Challenge Chamber, Vienna, Austria